CLINICAL TRIAL: NCT00653653
Title: Observational Study of the Pharmaco-Economic and Medical Effects of Optimising Medication Using Pharmacokinetic Pharmacogenomics and Medication Interaction Analysis in Private Practice.
Brief Title: Medication Optimisation for Reducing Events in a Private Practice Setting
Acronym: MORE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Awenydd GmbH (Industry)
Responsible Party: Dr. LS Griffith, awenydd Gene Diagnostic
Other Study IDs: AW_SH_08
Record Dates: First submitted 2008-04-02; First posted 2008-04-07 (Estimated); Last update posted 2009-04-08 (Estimated); Status verified 2009-04

CONDITIONS: Pharmacogenetic Analysis to Reduce Events.
Keywords: pharmacogenetics; pharmacoeconomics; adverse events; drug metabolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Group A: Recruited patients will be prospectively observed as one cohort with genotyping/medication interaction analysis after 3 months, followed up by a further 3 month observational period.

SUMMARY:
Using a prospective study design of two three month periods (before and after genotyping) in which the patients will self-monitor their health status and possible medical events it is hypothesized that it will be shown that patients having their medication altered to fit their genetic status and/or having their medication altered because of inherent interaction potential will have less recordable events after genotyping and medical analysis than before.

It is well known that ADRs (recordable adverse events to medication) are responsible for a large number of deaths and hospitalizations. Furthermore it is well recorded that genotyping of individual cytochrome P450 enzymes (2D6, 2C9, 2C19, among others) is directly related to a metabolic phenotype - fast metabolisers, slow metabolisers, intermediate and normal metabolisers. These differing phenotypes have altered metabolism of many medications and in a number of retrospective clinical trails it has been shown that ADRs and effect can be reduced/bettered through genotyping and alteration of medication.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years
* not demented
* 1 or more documented events in the previous 6 months.
* more than one medication
* multi-morbid

Exclusion Criteria:

* demented
* life expectancy less than 1 year
* heart attack within the last 6 months
* Marcumar® Therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-06 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
Reduction of reported events in the time frame. | 3 months

SECONDARY OUTCOMES:
Reduction of total costs associated per patient in the time frame. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Lee S Griffith, Ph.D., Study Director — Awenydd GmbH; André Gessner, MD Ph.D., Principal Investigator — University of Erlangen-Nürnberg
Locations (1):
- Awenydd Gmbh, Cologne, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Chialda L, Griffith LS, Heinig A, Pahl A. Prospective use of CYP pharmacogenetics and medication analysis to facilitate improved therapy - a pilot study. Per Med. 2008 Jan;5(1):37-45. doi: 10.2217/17410541.5.1.37. PMID 29783392